CLINICAL TRIAL: NCT02332343
Title: Sparing of the Fovea in Geographic Atrophy Progression
Acronym: SIGHT
Status: Completed | Type: Observational
Sponsor: University Hospital, Bonn (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Dr. Monika Fleckenstein, PD, Dr. med., University Hospital, Bonn
Other Study IDs: 173/14
Record Dates: First submitted 2015-01-04; First posted 2015-01-06 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Atrophy; Geographic Atrophy; Age-related Macular Degeneration; Eye Diseases
Keywords: Retina; Retinal pigment epithelium
MeSH Terms: conditions — Atrophy; Geographic Atrophy; Macular Degeneration; Eye Diseases

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No intervention - Natural history study

SUMMARY:
Dry age-related macular degeneration (AMD) is a common cause for severe visual loss in the elderly and represents an unmet need. So far no treatment is available for geographic atrophy (GA), which represents the advanced dry form characterized by expanding areas of outer retinal atrophy with corresponding absolute scotoma. The foveal retina may be spared until late in the course of the disease, a phenomenon termed "foveal sparing". However, the disease process ultimately also involves the central retina leading to irreversible loss of central vision. While the natural history of eyes with GA has been extensively studied with regard to the entire atrophic area, morphology-function analyses for "foveal sparing" GA in particular are still missing. Such data are needed for various purposes including the future use in interventional pharmacological trials aiming to slow the progression of GA and to preserve the foveal retina. In this study, different imaging modalities for accurate detection and quantification of preserved foveal retinal areas will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* The study eye must have a contiguous well-demarcated area of GA either in a complete ring around the spared fovea or in a horseshoe pattern with a total atrophy size of ≤ 7 Disk Areas
* Patient is willing to undergo ocular examination

Exclusion Criteria:

* The presence or history of CNV (choroidal neovascular membrane) in the study eye
* Ocular disease in the study eye that may confound assessment of the retina, other than non-exudative AMD (e.g., diabetic retinopathy, uveitis)
* Cataract surgery or ocular surgery in the study eye within 30 days prior to the baseline visit
* Current or previous participation in clinical studies investigating drugs, medical devices or supplements within 30 days prior to enrolment in the study - Previous or concomitant therapy to reat AMD (investigational or FDA approved); oral supplements of vitamins and minerals are permitted
* Known medical history of allergy or sensitivity to tropicamide or fluorescein dye that is clinically relevant in the investigator's opinion

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suitable for the study will be recruited at the University of Bonn, Department of Ophthalmology
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2014-10; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Best corrected visual acuity (BCVA) | baseline

SECONDARY OUTCOMES:
Size of Geographic atrophy area as determined by confocal laser scanning ophthalmoscopy (in mm²) | baseline
Size of foveal sparing area as determined by confocal laser scanning ophthalmoscopy (in mm²) | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Monika Fleckenstein, PD, Dr. med., Principal Investigator — University of Bonn
Locations (1):
- Department of Ophthalmology, University of Bonn, Bonn, North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Holz FG, Bindewald-Wittich A, Fleckenstein M, Dreyhaupt J, Scholl HP, Schmitz-Valckenberg S; FAM-Study Group. Progression of geographic atrophy and impact of fundus autofluorescence patterns in age-related macular degeneration. Am J Ophthalmol. 2007 Mar;143(3):463-72. doi: 10.1016/j.ajo.2006.11.041. Epub 2006 Dec 22. PMID 17239336
- [Background] Schmitz-Valckenberg S, Bultmann S, Dreyhaupt J, Bindewald A, Holz FG, Rohrschneider K. Fundus autofluorescence and fundus perimetry in the junctional zone of geographic atrophy in patients with age-related macular degeneration. Invest Ophthalmol Vis Sci. 2004 Dec;45(12):4470-6. doi: 10.1167/iovs.03-1311. PMID 15557456
- [Background] Schmitz-Valckenberg S, Fleckenstein M, Helb HM, Charbel Issa P, Scholl HP, Holz FG. In vivo imaging of foveal sparing in geographic atrophy secondary to age-related macular degeneration. Invest Ophthalmol Vis Sci. 2009 Aug;50(8):3915-21. doi: 10.1167/iovs.08-2484. Epub 2009 Apr 1. PMID 19339734
- [Derived] Lindner M, Pfau M, Czauderna J, Goerdt L, Schmitz-Valckenberg S, Holz FG, Fleckenstein M. Determinants of Reading Performance in Eyes with Foveal-Sparing Geographic Atrophy. Ophthalmol Retina. 2019 Mar;3(3):201-210. doi: 10.1016/j.oret.2018.11.005. Epub 2018 Nov 22. PMID 31014695